CLINICAL TRIAL: NCT05062122
Title: Evaluation of the Effects of Vibration and Kinesiology Tape Applications Applied to the Affected Side Forearm Extensor Muscles on Hand Skills in Children With Hemiplegic Cerebral Palsy
Brief Title: The Effects of Vibration and Kinesiology Tape Applications in Children With Hemiplegic Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Beyzanur Dikmen, physiotherapist, Kırıkkale University
Other Study IDs: kırıkkaleuniversity10
Record Dates: First submitted 2021-09-05; First posted 2021-09-30 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2022-09

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: cerebral palsy; kinesio tape; physiotherapy; vibration
MeSH Terms: conditions — Cerebral Palsy | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- vibration group: Vibration applied group in addition to conventional physiotherapy
  Interventions: Other: vibration group
- kinesiology tape group: The group in which kinesiology tape was applied in addition to conventional physiotherapy
  Interventions: Other: kinesiology tape group
- control group: Group receiving only conventional physiotherapy
  Interventions: Other: control group

INTERVENTIONS:
Other: vibration group — Hand skills were evaluated before and after 10 minutes of vibration application.
  Groups: vibration group
Other: kinesiology tape group — Dexterity was assessed before and after kinesiology tape application.
  Groups: kinesiology tape group
Other: control group — Manual dexterity was assessed before and after traditional physiotherapy.
  Groups: control group

SUMMARY:
The aim of this study was to evaluate the effects of vibration and kinesiology tape applications applied to the affected side forearm extensor muscles on dexterity in children with hemiplegic cerebral palsy.

DETAILED DESCRIPTION:
Upper extremity in children with hemiplegic cerebral palsy significantly more affected than the lower extremities. Child mostly does not use the affected side and activity and weight uses the solid side in the overlay. in the upper extremity One of the muscles most affected by spasticity is the wrist and wrist. finger flexors. Secondary in antagonist of these muscles weakness develops and posture disorders occur. In this study The kinesiology tape, which has been increasingly used in recent years, affected by the application and local vibration application. hand with application to the lateral forearm extensor muscle group comparing their effects on their skills with the control group. aimed to evaluate. As a result of the study, this diagnosis hand skills of which application in children who are studying has a greater effect on and in which rehabilitation that the application should be preferred more It will be a guide for physiotherapists.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hemiplegic cerebral palsy,
* No severe spasticity that prevents grasping and releasing an object (Modified which is at the level of 0, 1, 1+, 2 according to the Ashworth Scale),
* According to the Hand Skills Classification System (EBSS) at 1, 2 and 3 levels with function,
* Consisting of children between the ages of 4-18,
* Being treated in a special education and rehabilitation center,
* The family accepts the participation of their child in the study.
* They are children who have the mental level to take basic commands.

Exclusion Criteria:

* Having severe mental retardation that prevents communication and taking basic commands,
* The family does not accept the child to work,
* Severe spasticity that prevents grasping an object (Modified Ashworth 3 and 4 levels according to the scale),
* Hand function at 4 and 5 levels according to the Hand Skills Classification System (EBSS) the one which,
* Compliance and behavior during the application of the tests used to obtain the data are children with the disorder.

Ages: 4 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Able to take basic commands between the ages of 4 and 18
  1, 2, 3 according to the Manual Ability Classification System Children with hemiplegic cerebral palsy with a value of 0, 1, 1+, 2 on the Modified Ashworth Scale
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Nine Hole Peg Test (DDPT) | 10 months
  DDPT is a standard-sized nine-hole panel. Nine nails made of simple, performance-enhancing material is a time-tested test of fine upper motor function. To counter the learning effect, the child was allowed to experience this test. Before the start of the test, the test procedure is explained as quickly as possible. After inserting wooden nails into the holes in the same way and placing all 9 nails into the holes, the nails were asked to be removed without waiting. Test completion time recorded with the stopwatch. The stopwatch was stopped when the last nail was removed and placed in the side chamber, and the time displayed on the stopwatch was recorded. The completion time of the test gave information about the person's upper extremity performance.
Wooden Box and Block Test (TKBT) | 10 months
  CBCT is used to evaluate manual dexterity in patients with stroke, multiple sclerosis, traumatic brain injury, fibromyalgia, children with upper extremity involvement, and the elderly. While the test is seated in a chair with a backrest without armrests, supported by the feet, the affected side to be evaluated is conventionally positioned with the hand. It was performed before and after the application in addition to physiotherapy. First, a trial period of 15 seconds was given. Then, he was asked to fill 150 small wooden blocks one by one as fast as possible for 60 seconds from the box with the hand to be tested to the box next to it. If he throws it without raising his hand, it will not be counted, accidentally 2 It was stated that if he throws a wooden block, it will be counted as 1 wooden block. It was counted how many wooden blocks were thrown in 60 seconds and the result gave information about the upper extremity performance tested.

SECONDARY OUTCOMES:
Manual Skills Classification System (EBSS) | 10 months
  The EBSS was a five-level, ordinal classification system that described the manual dexterity of children with CP aged 4 to 18 years when handling objects in typical daily activities. EBSS levels define the use of both hands in daily activities, which is expected according to a child's age, not only as a fine motor function, but also as dependent on cognitive, motor planning and motivation. EBSS is not an outcome measure or diagnostic tool, its purpose is a child's daily classifying the ability to use objects manually in life. EBSS level 1 represents the highest level of manual ability at which objects can be grasped and used easily and successfully, and level 5 represents the lowest level where objects cannot be used independently and assistance is most needed.
Modified Ashworth Scale (MAS) | 10 months
  The MAS is the most universally accepted clinical tool used to measure the increase in muscle tone. In 1964, Bryan Ashworth published the Ashworth Scale as a method of grading spasticity while working with multiple sclerosis patients. The original Ashworth scale was 0-4, 0 without resistance, and 4 for spasticity. It is a 5-point numerical scale with limb stiffness in flexion or extension. In 1987, manual testing of elbow flexor muscle spasticity, Bohannon and Smith, while conducting a study to examine inter-interpretive reliability, modified the Ashworth scale to add 1+ to the scale to increase sensitivity. The purpose of the modified Ashworth scale is to assess muscle tone. It is easy to use, but the findings are subject to the subjective opinion of the evaluator. This scale classifies muscle tone from 0 (normal) to 4 (severe spasticity).
ABILHAND-Kids Manual Ability Scale | 10 months
  ABILHAND Kids, developed by Rasch in 2004, is a reliable, valid and sensitive measure for assessing manual dexterity in children with upper extremity disorders. ABILHAND-Kids is a convenient and fast-applied scale consisting of 21 items covering various areas of daily life. Often the function of both hands is evaluated. Generally, the scale is applied by asking the families, if the child is older and at a level to be able to apply the scale, he/she can be included in the application. While assessing functional ability, any assistive device or There should be no human support. For each item, they are asked to indicate their perceived difficulty on a three-level scale: Impossible (0 point), Difficult (1 point), or Easy (2 points).

CONTACTS AND LOCATIONS:
Overall Officials: Beyzanur Dikmen, Study Director — Graduate student at Kırıkkale University; Meral Sertel, Study Chair — Associate professor at Kırıkkale University
Locations (1):
- Private Karma Special Education and Rehabilitation Center, Ankara, Turkey (Türkiye)